CLINICAL TRIAL: NCT01499329
Title: Endovascular Treatment of Iliac Artery Occlusions or Stenoses Using the Zeus CC Stent System
Brief Title: Safety and Performance of the Zeus CC Stent for the Treatment of Iliac Occlusive Disease
Acronym: EAZY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: be Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-EAZY-05-002
Record Dates: First submitted 2011-10-11; First posted 2011-12-26 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Peripheral Artery Disease
Keywords: Stent therapy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient receiving stent therapy

SUMMARY:
The purpose of this study is to evaluate safety and performance of the balloon-expandable Zeus CC (Rontis AG) stent for the treatment of Trans-Atlantic Inter-Society Consensus (TASC) A, B, C and D iliac lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is older than 18 years
2. Patient must sign a written informed consent form that is approved by the ethics committee prior to index-procedure
3. Patient must be compliant with all follow-up visits
4. Patient suffers from intermittent claudication (Rutherford 1-3) or critical limb ischemia (Rutherford 4 and 5)
5. Patient's life expectancy is more than 2 years
6. Patient has iliac atherosclerotic de novo lesion(s) type A, B, C & D according to TASC-II classification
7. Target vessel diameter is between 5 and 9 mm
8. Target lesion has a baseline diameter stenosis of more than 50%
9. Patient has sufficient infra-inguinal run-off with at least a patent common femoral artery and deep femoral artery (both <50% stenosis)

Exclusion Criteria:

1. Patient has a life expectancy of less than 2 years
2. Patient is refusing to be compliant with all follow-up visits
3. Patient suffers from acute limb ischemia, defined as any sudden decrease in limb perfusion causing a potential threat to limb viability.
4. Patient is intolerant to anticoagulant or antiplatelet therapy such as aspirin, heparin, clopidogrel or ticlopidine drug therapy
5. Patient has already been treated with a stent in the ipsilateral target vessel
6. Patient suffered tissue loss in the target extremities, defined as Rutherford 6
7. Patient is already enrolled in this or another investigational device study
8. Patient had a coronary intervention within the last 60 days before enrolment into this study or there is a planned coronary intervention within 60 days of enrolment into this study
9. Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index-procedure
10. Any planned surgical intervention within 30 days of the index-procedure
11. Patient has an abdominal aortic aneurysm that is likely to require repair within the next 2 years.
12. Patient has no sufficient infra-inguinal run-off (>50% stenosis). Patient inclusion is only possible if revascularization (endovascular or surgical) is performed in the same procedure with a peroperative angiographic control yielding <30% stenosis.
13. Target lesion is a restenotic lesion.
14. Target lesion is adjacent an aneurysm.
15. Target vessel perforation with documented contrast extravasation during index-procedure prior to stent placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iliac occlusive disease TASC A, B, C and D lesions.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Binary (≥ 50%) restenosis rate | 12, 24 months
  assessed by duplex ultrasound at the target lesion without the need for repeat TLR after the index-procedure in surviving patients with preserved limbs

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Letter, MD, Principal Investigator — AZ Sint Jan Bruges
Locations (1):
- AZ Sint Jan Bruges, Bruges, Belgium